CLINICAL TRIAL: NCT05341518
Title: Subscapularis Repair During Reverse Total Shoulder Arthroplasty: a Randomized Control Trial
Brief Title: Subscapularis Repair During Reverse Total Shoulder Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Participating sites failed to secure funding and study was not feasible at one site.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Guido Marra, Professor of Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00215591
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Shoulder Osteoarthritis; Arthropathy Shoulder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subscapularis repair (Experimental): Patients will undergo standard of care reverse total shoulder arthroplasty with subscapularis repair
  Interventions: Procedure: Subscapularis repair
- No repair (No Intervention): Patients will undergo standard of care reverse total shoulder arthroplasty. The subscapularis will not be repaired.

INTERVENTIONS:
Procedure: Subscapularis repair — To complete reverse total shoulder arthroplasty, the surgeon must cut through the subscapularis muscle. In this arm of the study, the muscle will be repaired, rather than left to heal itself.
  Arms: Subscapularis repair

SUMMARY:
This multi-site study involving Northwestern Medicine, Beaumont Health, and Loyola Medicine seeks to answer the following question: do patients who undergo subscapularis (SSc) repair during reverse total shoulder arthroplasty (RSA) have better post-operative outcomes than patients who do not undergo SSc repair during RSA? The investigators hypothesize that patients who do not undergo SSc repair during RSA have better post-operative outcomes than patients who undergo SSc repair during RSA. This study will address the controversy surrounding SSc repair during RSA via a multi-institutional randomized controlled trial that will compare clinical outcomes of patients who receive SSc repair during RSA to those who do not.

ELIGIBILITY:
Inclusion Criteria:

1. Primary RSA procedure with repairable (intact) SSc
2. Operation will be performed by a participating surgeon using Zimmer Biomet Comprehensive Reverse Shoulder System implant
3. Diagnosis with imaging of arthropathy with rotator cuff insufficiency
4. Surgical approach: Deltopectoral
5. Fluent English speakers/readers

Exclusion Criteria:

1. Minor (<18 y/o)/vulnerable populations (pregnant women, prisoners, adults unable to consent)
2. Revision surgery
3. Oncologic surgery
4. non-ZB CRSS implants
5. Unrepairable SSc

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The American Shoulder and Elbow Surgeons (ASES) Shoulder Score | up to 12 months post-surgery
  Scored from 0 (worst shoulder condition) to 100 (best shoulder condition)

SECONDARY OUTCOMES:
Internal Rotator (IR) Strength | up to 12 months post-surgery
  IR at the side and supported IR at 90˚ scapation; percent of nonsurgical side
PROMIS Bank v1.1 - Pain Interference | up to 12 months post-surgery
  PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population (usually U.S. general population).
Shoulder Range of Motion | up to 12 months post-surgery
  shoulder extension, flexion, internal rotation, abduction, adduction; percent of nonsurgical side

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marra, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (2):
- United States (2):
  - Loyola Medicine, Maywood, Illinois
  - Beaumont Health, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No
There is no participant data to share. No participants were enrolled.